CLINICAL TRIAL: NCT02813122
Title: The Use of X-ray in Bariatric Surgeries
Status: Completed | Type: Observational
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Sergio Gabriel Susmallian, Head of Surgery department, Assuta Medical Center
Other Study IDs: 0016-16-ASMC
Record Dates: First submitted 2016-06-19; First posted 2016-06-24 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Complications of Bariatric Procedures; X-rays; Effects
MeSH Terms: interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- with x-ray: patients underwent bariatric surgery and underwent x-ray
  Interventions: Device: x-ray
- without x-ray: patients underwent bariatric surgery and did not underwent x-ray

INTERVENTIONS:
Device: x-ray — x-ray for the detection of leaks and bleeding
  Groups: with x-ray

SUMMARY:
examination of the importance of the use of X-ray in bariatric surgery outcome.

DETAILED DESCRIPTION:
the x-ray will be used in order to evaluate the number of complications occured during bariatric surgeries such as bleeding, leak, etc. a retrospective analysis of patients with those complications will be performed and the presence of the x-ray and its findings will also be documented.

ELIGIBILITY:
Inclusion Criteria:

first bariatric surgery

Exclusion Criteria:

recurrent bariatric surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients underwent bariatric surgery between 2011-2015
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Actual)
Dates: Start 2016-06; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
complications | retrospective- data collection and analysis will be ended in six months.
  the outcome measure will be assessed and data will be presented in six months

CONTACTS AND LOCATIONS:
Overall Officials: Sergio G Susmallian, M.D, Principal Investigator — Assuta Medical Center
Locations (1):
- Assuta Medical Center, Tel Aviv, Israel, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Susmallian S, Folb E, Barnea R, Raziel A. Comparison of Imaging Modalities for Detecting Complications in Bariatric Surgery. Obes Surg. 2018 Apr;28(4):1063-1069. doi: 10.1007/s11695-017-2970-5. PMID 29047049